CLINICAL TRIAL: NCT06136923
Title: An Exploratory Study to Evaluate Attention Biases in Adults With Multiple Sclerosis, Breast Cancer, and Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CT-100-D-004
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Lung Cancer; Breast Cancer
Keywords: Prescription digital therapeutic (PDT); Software as a Medical Device (SaMD); Smartphone app; Attention Biases; Cognition; Multiple Sclerosis; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Multiple Sclerosis; Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Multiple Sclerosis with Mobility Limitations Study App A (Experimental): Cognitive Training App CT-100-D-004-A uses implicit training with audiovisual stimuli to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for multiple sclerosis with mobility limitations.
  Interventions: Device: CT-100-D-004-A
- Multiple Sclerosis with Mobility Limitations Study App B (Other): Cognitive Training App CT-100-D-004-B uses implicit training with verbal processing exercises to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for multiple sclerosis with mobility limitations.
  Interventions: Device: CT-100-D-004-B
- Multiple Sclerosis without Mobility Limitations Study App A (Experimental): Cognitive Training App CT-100-D-004-A uses implicit training with audiovisual stimuli to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for multiple sclerosis without mobility limitations.
  Interventions: Device: CT-100-D-004-A
- Multiple Sclerosis without Mobility Limitations Study App B (Other): Cognitive Training App CT-100-D-004-B uses implicit training with verbal processing exercises to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for multiple sclerosis without mobility limitations.
  Interventions: Device: CT-100-D-004-B
- Oncology Breast Cancer Study App A (Experimental): Cognitive Training App CT-100-D-004-A uses implicit training with audiovisual stimuli to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for breast cancer.
  Interventions: Device: CT-100-D-004-A
- Oncology Breast Cancer Study App B (Other): Cognitive Training App CT-100-D-004-B uses implicit training with verbal processing exercises to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for breast cancer.
  Interventions: Device: CT-100-D-004-B
- Oncology Lung Cancer Study App A (Experimental): Cognitive Training App CT-100-D-004-A uses implicit training with audiovisual stimuli to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for lung cancer.
  Interventions: Device: CT-100-D-004-A
- Oncology Lung Cancer Study App B (Other): Cognitive Training App CT-100-D-004-B uses implicit training with verbal processing exercises to potentially redirect and modulate attention processes. This intervention is designed to help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli for lung cancer.
  Interventions: Device: CT-100-D-004-B

INTERVENTIONS:
Device: CT-100-D-004-A — Attention Biases App CT-100-D-004-A Digital Neuro-activation and Modulation (DiNaMo) component uses implicit training to redirect and strengthen attention processes. This intervention can help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli.
  Arms: Multiple Sclerosis with Mobility Limitations Study App A; Multiple Sclerosis without Mobility Limitations Study App A; Oncology Breast Cancer Study App A; Oncology Lung Cancer Study App A
Device: CT-100-D-004-B — Attention Biases App CT-100-D-004-B Digital Neuro-activation and Modulation (DiNaMo) component uses implicit training to redirect and strengthen attention processes. This intervention can help improve cognitive capabilities as well as redirect attentional biases to make participants less sensitive to distressing stimuli.
  Arms: Multiple Sclerosis with Mobility Limitations Study App B; Multiple Sclerosis without Mobility Limitations Study App B; Oncology Breast Cancer Study App B; Oncology Lung Cancer Study App B

SUMMARY:
CT-100 is a platform that provides interactive, software based therapeutic components that may be used as part of a treatment in future software-based prescription digital therapeutics. One class of CT-100 components are Digital Neuro-activation and Modulation (DiNaMo) components. DiNaMo components target key neural systems (including but not limited to systems related to sensory-, perceptual-, affective-, pain-, attention-, cognitive control, social- and self-processing) to optimally improve a participant's health.

DETAILED DESCRIPTION:
CT-100 is a platform that provides interactive, software based therapeutic components that may be used as part of a treatment in future software-based prescription digital therapeutics. One class of CT-100 components are Digital Neuro-activation and Modulation (DiNaMo) components. DiNaMo components target key neural systems (including but not limited to systems related to sensory-, perceptual-, affective-, pain-, attention-, cognitive control, social- and self-processing) to optimally improve a participant's health.

Targeted cognitive training is used to reduce symptoms relevant to multiple sclerosis (MS) and cancer. Biases to direct attention towards or away from certain stimuli can exacerbate a variety of symptoms in many different indications. For example, in chronic pain conditions, patients are more attentive to pain-related stimuli, which can lead to hypersensitization. Similarly, hypersensitivity to threat-related stimuli can exacerbate anxiety.

In this treatment, users are trained to re-orient attention away from negative stimuli, such as pain- or threat-related stimuli.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be eligible for entry into the study if all of the following criteria are met:

  1. Fluent in written and spoken English, confirmed by ability to read, understand, and sign the informed consent form
  2. Lives in the United States
  3. Adult between 22 and 65 years old
  4. Meets indication-specific including criteria, as reported by the study participant with adequate clinical documentation (to be provided to the study team upon request)
  5. Has an active email address and is willing and able to receive and respond to email messages
  6. Has access to an internet connection during the study duration
  7. Has an active PayPal account to receive study compensation, or is willing to create one
  8. Willing and able to comply with study protocol and assessments
  9. Is the sole user of an iPhone with an iPhone operating system (iOS) version 14 or later or a smartphone with an Android operating system (OS) version 10 or later for the duration of the study
  10. Is willing and able to receive Short Message Service (SMS) text messages and notifications on their smartphone
  11. Has access to operating headphones

Exclusion Criteria:

* A participant will not be eligible for study entry if any of the following criteria are met:

  1. Visual, dexterity or cognitive deficit so severe that it precludes the use of an App-based reaction time-based activity per investigator judgment
  2. Severe psychiatric disorder involving a history of psychosis (e.g., schizophrenia, bipolar disorder, severe personality disorders)
  3. Psychiatric hospitalization in the past 6 months
  4. Participation in any research study (including studies on psychotherapy, mindfulness, cognitive training or pharmacological treatment) during the past 3 months
  5. Initiation or change in primary disease-specific medication within 30 days prior to entering the study
  6. Planning the introduction of new therapies (including studies on psychotherapy, mindfulness, cognitive training or pharmacological treatment) during the study duration (6 weeks)
  7. Anticipating a change in current pharmacological or psychotherapy treatment regimen during the study period (6 weeks)
  8. Self-reported substance use disorder within the past 1 year
  9. Severe neurological disorders impairing brain function (e.g., previous stroke, dementia, primary brain function, brain metastases, Alzheimer's disease, Parkinson's disease, history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities)
  10. Mild, moderate, severe or profound unilateral or bilateral hearing loss

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Change in Patient Reported Outcomes | Baseline to Week 4
  Change from baseline to Week 4 in quality of life as measured by PROMIS-29+2 (Patient Reported Outcomes Measurement Information System)

SECONDARY OUTCOMES:
Change in Pain Severity and Pain Interference | Baseline to Week 4
  Change from baseline to Week 4 in pain severity and pain interference as measured by the Brief Pain Inventory (BPI)
Change in Pain Catastrophizing Scale | Baseline to Week 4
  Change from baseline to Week 4 Pain Catastrophizing Scale (PCS) from 0-30+
Change in indication-specific measures MS | Baseline to Week 4
  Change from baseline to Week 4 in indication-specific measures: Symbol Digit Modalities Test (SDMT) for MS
Change in indication-specific measures Cancer | Baseline to Week 4
  Change from baseline to Week 4 in indication-specific measures: Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) for cancer
Proportion of participants with an improvement | Baseline to Week 4
  Proportion of participants with an improvement as measured by the Global Rating of Change (GRC) score from -5 to 5 at Week 4
Engagement with Study App | Baseline to Week 4
  Engagement with the Study App as measured by daily time in the Study App

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States